CLINICAL TRIAL: NCT02349191
Title: A Prospective, Single Site, Single Arm, Non-randomized, Interventional Study to Evaluate the Safety and Effectiveness of Omental Transposition Surgery for Patients With Alzheimer's Disease.
Brief Title: Omental Transposition Surgery for Mild Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bariatric Medicine Institute, Salt Lake City, UT (Other)
Responsible Party: Principal Investigator, Dr. Daniel Cottam, Director Bariatric Medicine Institute, Bariatric Medicine Institute, Salt Lake City, UT
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cottam - 1
Record Dates: First submitted 2015-01-12; First posted 2015-01-28 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimers; dementia; omental transposition; neurological
MeSH Terms: conditions — Alzheimer Disease; Dementia; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional cohort (Experimental): Omental transposition for mild Alzheimers Disease
  Interventions: Procedure: Omental transposition for mild Alzheimers disease

INTERVENTIONS:
Procedure: Omental transposition for mild Alzheimers disease — An omental pedicle is brought from the abdomen underneath the skin and sewn to the dura matter of the brain via a craniotomy.

SUMMARY:
This study is a prospective, single arm, non-randomized, interventional study to evaluate the safety and effectiveness of Omental transposition (OT) in subjects with early stage AD.

Within-subjects (repeated-measures) design will be utilized to compare follow-up outcomes to baseline.

The following assessments will be performed at baseline, then at 1, 3, 6, 12, and 24 months following surgery:

* Montreal Cognitive Assessment (MoCA)
* Alzheimer's Disease Assessment Scale-Cognition (ADAS-Cog)
* General Practitioner Assessment of Cognition (GPCOG)
* Eight-item Informant Interview to Differentiate Aging and Dementia (AD8) Subjects who have early stage AD confirmed by a neuropsychological test (MoCA) and who are healthy enough to undergo surgery.

The experimental procedure to be performed is omental transposition (OT) surgery. It will be performed as a laparoscopic or open procedure for omental lengthening and an open procedure for brain access, with a general surgeon performing the omental lengthening/tunneling and a neurosurgeon performing brain access/brain biopsy/omental placement on brain.

Up to twenty-five (25) subjects, with the first 5 subjects being part of a learning curve group and the next 20 subjects being part of the experimental group.

The duration of each subject's participation will be approximately 25 months from screening through the 24 month follow-up visit.

DETAILED DESCRIPTION:
The experimental procedure to be performed is omental transposition surgery, during which a general surgeon and a neurosurgeon work as a team to transpose a pedicle omental graft to the surface of the brain. The general surgeon is responsible for performing a laparotomy/laparoscopy, elongating the omentum into a long pedicle and developing an extensive subcutaneous tunnel up the chest and neck to the head. The neurosurgeon is responsible for performing the craniotomy and securing the omentum on the brain.

Creating an intact omental pedicled flap requires the services of a general surgeon and neurosurgeon. The first step in the operation is to obtain access to the abdominal cavity laparoscopically using four 5cm trocars, or via laparotomy through an upper midline incision. The omentum is then removed from the transverse colon, after which it is separated from its proximal and central attachments to the stomach. The omentum detachments are made directly on the greater curvature of the stomach, leaving the gastroepiploic arteries and veins within the still-connected omentum apron.

Final separation of the omentum from the proximal portion of the stomach is done by dividing the left gastroepiploic vessels, which at the highest proximal level on the stomach become the short gastric vessels. The vascular connections to and from the omentum are now maintained solely from the right gastric and right gastroepiploic vessels. In order for the omental pedicle graft to reach the brain without tension, further surgical tailoring of the omentum is carried out, with care being taken to ensure the preservation of a major omental artery and vein.

After the omentum has been lengthened to an appropriate extent to reach the head, several small (3- to 4-inch) transverse incisions are made on the chest wall slightly lateral to the midline, with the side of the midline to make the transverse incisions depending on which cerebral hemisphere the omentum is to be placed. These transverse incisions are connected subcutaneously, thus creating a tunnel that begins at the upper pole of the midline abdominal incision and travels subcutaneously, up the chest wall and neck to behind the ear.

Although the subcutaneous tissue behind the ear is extremely dense, it is essential that the tunnel at this location be at least 2-3 finger lengths in width so that there is no constriction on the omentum in this particular area within the tunnel. As the omentum in the tunnel passes behind the ear, it goes beneath the base of the scalp flap that had been previously dissected in making the initial craniotomy incision.

The neurosurgery portion of the operation involves removal of a single piece of bone over the temporal-frontal area, opening the dura mater, followed by the removal of patches of arachnoid membrane, with care being taken to avoid blood vessels on the surface of the brain.

At this point in the operation, the omentum is laid directly upon the parietal-temporal-frontal area, after which the dura mater is sutured to the omentum. It is not necessary that the edges of the omentum be applied to the cut edges of the dura since the omentum can be tucked under the edges of the dura for greater coverage of the brain. The edges of the dura are then sewn to the top surface of the omentum using absorbable sutures and the craniotomy is closed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 60 to 85 years of age
2. Montreal Cognitive Assessment (MoCA) score of 11 to 18 (mild AD)
3. Healthy enough to undergo the surgical procedure based on surgical risk factor definitions (ASA ≤ 3, using the ASA classification)
4. Must be able to read and understand English in order to complete all AD assessments
5. All medical illnesses other than dementia must be well controlled
6. Must have legally authorized caregiver if incapable of making their own decisions who is willing and able to perform the following:

   1. provide informed consent if the subject is unable to do so;
   2. monitor the subject;
   3. answer informant based questionnaires;
   4. provide transportation and accompany the subject to all visits
7. Subject or caregiver is willing and able to provide written informed consent and assent (if applicable)
8. Subject and/or caregiver are willing to comply with the study procedures and complete the entire study as specified in the protocol

Exclusion Criteria:

1. Life expectancy < 2 years
2. Subject who had or has cancer and is undergoing cancer therapy
3. Previous course of abdominal, cranial or neck radiotherapy or chemotherapy
4. Patients with neck calcifications may be excluded
5. Subject with uncontrolled heart disease, renal disease, or liver disease
6. Subject with diabetes mellitus whose glycoslated Hb (A1C) > 7
7. Complete blood count (CBC) with white blood cell <4,000 or platelets >125,000
8. Subject with uncontrollable hypertension (HTN)
9. Subject with previous abdominal surgery or disorder that could negatively influence the outcome of the OT surgery
10. Subject who has had a craniotomy in the past
11. Recent major surgery within the past 6 months
12. Use of cholinesterase inhibitors within the last 30 days and inability to not take cholinesterase inhibitors throughout the length of the study (about 25 mos)
13. Subject uses non-prescribed drugs of abuse or has a history of drug or alcohol abuse/dependence
14. Use of anticoagulants other then anti-platelet medications
15. Subject has significant central nervous system (CNS) disorder other than Alzheimer's disease
16. Subject has clinical evidence or history of stroke, transient ischemic attack, significant head injury or other unexplained or recurrent loss of consciousness ≥15 minutes
17. Major depressive disorder, schizophrenia, other psychotic disorders, or bipolar disorder
18. Subject has epilepsy
19. Patients with severe extra pyramidal signs
20. Patients with plastic surgery of the neck or face
21. Subject resides in hospital or moderate to high dependency continuous care facility
22. Non-English speaking subjects and/or caregivers
23. Subject has any condition that, in the opinion of the Investigator would preclude the use of the study procedure, may interfere with the evaluation of the procedure-related outcomes, or preclude the subject from completing the follow-up requirements

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-04 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical complications from beginning of anesthesia to discharge from Intensive Care Unit. | Participants will be monitored for postoperative complications for the duration of their hospital stay, an expected average of 2 days.
  surgical complications will be assessed from the anesthesia start time through hospital discharge.Total incidence (%) of complications will be calculated and reported,using Clavien-Dindo Classification of Surgical Complications.

SECONDARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale - Cognition (ADAS-cog) score from baseline at 12 months. | 12 months
  Percentage of score change, compared to baseline
Change in Montreal Cognitive Assessment (MoCA) score from baseline at 12 months | 12 months
  Percentage of score change, compared to baseline
Change in General Practitioner Assessment of Cognition (GPCOG) score from baseline at 12 months | 12 months
  Percentage of score change, compared to baseline
Change in Eight-item Informant Interview to Differentiate Aging and Dementia (AD8) score from baseline at 12 months | 12 months
  Percentage of score change, compared to baseline
Change in Alzheimer's Disease Assessment Scale - Cognition (ADAS-cog) score from baseline at 24 months | 24 months
  Percentage of score change, compared to baseline
Change in Montreal Cognitive Assessment (MoCA) score from baseline at 24 months | 24 months
  Percentage of score change, compared to baseline
Change in General Practitioner Assessment of Cognition (GPCOG) score from baseline at 24 months | 24 months
  Percentage of score change, compared to baseline
Change in Eight-item Informant Interview to Differentiate Aging and Dementia (AD8) score from baseline at 24 months | 24 months
  Percentage of score change, compared to baseline

REFERENCES:
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Goldsmith HS. Omental transposition for Alzheimer 's disease. Neurol Res. 1996 Apr;18(2):103-8. doi: 10.1080/01616412.1996.11740387. PMID 9162863
- [Background] Goldsmith HS. Treatment of Alzheimer's disease by transposition of the omentum. Ann N Y Acad Sci. 2002 Nov;977:454-67. doi: 10.1111/j.1749-6632.2002.tb04851.x. PMID 12480786
- [Background] Goldsmith HS. Omental transposition in treatment of Alzheimer disease. J Am Coll Surg. 2007 Dec;205(6):800-4. doi: 10.1016/j.jamcollsurg.2007.06.294. Epub 2007 Sep 18. No abstract available. PMID 18035264
- [Background] Goldsmith HS, Sax DS. Omental transposition for cerebral infarction: a 13-year follow-up study. Surg Neurol. 1999 Mar;51(3):342-5; discussion 345-6. doi: 10.1016/s0090-3019(98)00098-6. PMID 10086501
- [Background] Shankle WR, Hara J, Bjornsen L, Gade GF, Leport PC, Ali MB, Kim J, Raimo M, Reyes L, Amen D, Rudy L, O'Heany T. Omentum transposition surgery for patients with Alzheimer's disease: a case series. Neurol Res. 2008 Apr;30(3):313-25. doi: 10.1179/016164107X230126. Epub 2007 Aug 31. PMID 17767812
- See also: The Omentum — http://link.springer.com/chapter/10.1007/978-1-4612-3436-4_4